CLINICAL TRIAL: NCT03708653
Title: Association Between Some Candidate Single Nucleotide Polymorphisms and Postherpetic Neuralgia
Brief Title: Single Nucleotide Polymorphisms (SNPs) Associated With Postherpetic Neuralgia
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0904
Record Dates: First submitted 2018-09-05; First posted 2018-10-17 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2018-09

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHN(+): Patients who have persistent pain more than three months after the onset of herpes zoster.
- PHN(-): Patients whose pain disappear within three months.

SUMMARY:
Postherpetic neuralgia (PHN) is a common condition and affecting 5 to 30% of the herpes zoster patients. In some cases, the pain remained refractory after first and second line treatment for herpes zoster. This suggests that there may be genetic variants that make some patients susceptible to PHN. Using saliva samples from herpes zoster patients the investigators are going to analyze the relationship between single nucleotide polymorphisms (SNPs) in genes that are known to be involved in pain and PHN.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 50 years
* Clinically defined herpes zoster patients

Exclusion Criteria:

* Patients not able to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Herpes zoster patients in a large university hospital
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
correlation between pain SNPs and PHN | At Enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Director — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China